CLINICAL TRIAL: NCT05509647
Title: Unfractionated Heparin in COVID-19 and Non-COVID-19 Patients - an Observational Study.
Brief Title: Unfractionated Heparin in COVID-19 and Non-COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, edejonge, Head of the Intensive Care Department, Leiden University Medical Center
Other Study IDs: CoCo 2022-020
Record Dates: First submitted 2022-04-25; First posted 2022-08-22 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Heparin Overdose of Undetermined Intent; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Heparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 patients: Adult patients treated with unfractionated heparin aiming at aPTT 60-80 sec and/or anti-Xa level 0.3-0.7 iE/ml. All patients have Covid-19 proven by PCR or nose- or airway swab. Patients admitted to the ICU from the 15th of March 2020 until January 2022.
  Interventions: Drug: Unfractionated heparin
- non-COVID-19 patients: Adult patients treated with unfractionated heparin aiming at aPTT 60-80 sec and/or anti-Xa level 0.3-0.7 iE/ml. Patients admitted to the ICU between the 1st of January 2014 and the 1st of January 2020 are included.
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Unfractionated heparin — Patients are treated with unfractionated heparin aiming at aPTT 60-80 sec and/or anti-Xa levels of 0.3-0.7 iE/ml

SUMMARY:
The majority of ICU patients with COVID-19 show profound activation of coagulation, potentially resulting in thromboembolic events. In the treatment of these thromboembolic events it seemed that very high dosages of unfractionated heparin were necessary to achieve therapeutic values of aPTT and anti-Xa levels. The aim of this study is to explore whether heparin dosages are higher in COVID-19 patients compared to non-COVID-19 patients, to determine the correlation between aPTT and anti-Xa values and to explore possible causes for non-correlating aPTT and anti-Xa, including CRP and AT plasma levels.

DETAILED DESCRIPTION:
CoVID-19 is a viral disease caused by SARS-CoV-2 virus that may affect many organ systems. Patients with severe disease almost invariably have profound pulmonary inflammation and may require mechanical ventilation and prolonged ICU admission. Mortality in ICU patients may be up to 50%. In the majority of patients with CoVID-19 in the ICU, profound activation of coagulation is present as reflected by d-dimer levels up to 20.000 mg/L or higher. Patients with proven pulmonary thrombosis are commonly treated with unfractionated heparin (UFH). Typically, it seemed that very high dosages of UFH were necessary to achieve therapeutic values of aPTT and anti-Xa levels in COVID-19 patients. Though, the question remains whether dosages given in COVID-19 patients were indeed extravagant compared to non-COVID-19 patients and what potential causes of these high dosages might be. Earlier research already implied that APTT, which is a primarily used parameter to dose UFH, is not accurate and rather anti-Xa levels should be used. Other potential reasons for the high doses are that COVID-19 patients show signs of heparin resistance, possible due to high inflammation parameters. As overdosing of heparin can lead to serious bleeding complications, more understanding on heparin dosage, e.g. parameters to rely on and potential influencing factors, in COVID-19 patients is needed. The primary objective of this study is to determine whether heparin dosages are higher in COVID-19 patients compared to non COVID-19 patients. The secondary objective is to determine the correlation between aPTT and anti-Xa values and to explore possible causes for non-correlating aPTT and anti-Xa, including CRP and AT plasma levels.

ELIGIBILITY:
Inclusion Criteria Covid-19 group:

* Covid-19 disease proven by PCR of nose- or airway sample
* Age ≥ 18 years
* Admitted to the ICU from the 15th of March 2020 until 1st of January 2022
* Treated with unfractionated heparin aiming at aPTT 60-80 sec and/or anti-Xa level 0.3-0.7 iE/ml

Inclusion Criteria non-Covid-19 group:

* Age ≥ 18 years
* Admitted to the ICU between the 1st of January 2014 and 1st of January 2020
* Treated with unfractionated heparin aiming at aPTT 60-80 sec and/or anti-Xa level 0.3-0.7 iE/ml

Exclusion Criteria:

- Treatment with anticoagulants other than UFH or fibrinolytics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU in the above mentioned periods of time and in need for unfractionated heparin treatment are eligible to participate in the study. There is no selection bias: all patients fulfilling the entry criteria will be included.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Heparin dosage | Until end of heparin therapy or ICU discharge, whatever comes first.
  To determine whether heparin dosages are higher in COVID-19 patients compared to non COVID-19 patients.

SECONDARY OUTCOMES:
Correlation between aPTT and anti-Xa values | Until end of heparin therapy or ICU discharge, whatever comes first.
  To explore possible causes for non-correlating aPTT and Anti-Xa levels
Correlation between non-correlating aPTT and Anti-Xa levels and CRP | Until end of heparin therapy or ICU discharge, whatever comes first.
  To explore possible causes for non-correlating aPTT and Anti-Xa levels
Correlation between non-correlating aPTT and Anti-Xa levels and AT plasma levels | Until end of heparin therapy or ICU discharge, whatever comes first.
  To explore possible causes for non-correlating aPTT and Anti-Xa levels

CONTACTS AND LOCATIONS:
Overall Officials: Evert de Jonge, MD, PhD, Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Thachil J, Tang N, Gando S, Falanga A, Levi M, Clark C, Iba T, Cattaneo M. Type and dose of heparin in Covid-19: Reply. J Thromb Haemost. 2020 Aug;18(8):2063-2064. doi: 10.1111/jth.14870. Epub 2020 May 11. No abstract available. PMID 32329221
- [Background] Arachchillage DRJ, Kamani F, Deplano S, Banya W, Laffan M. Should we abandon the APTT for monitoring unfractionated heparin? Thromb Res. 2017 Sep;157:157-161. doi: 10.1016/j.thromres.2017.07.006. Epub 2017 Jul 6. PMID 28759760
- [Background] White D, MacDonald S, Bull T, Hayman M, de Monteverde-Robb R, Sapsford D, Lavinio A, Varley J, Johnston A, Besser M, Thomas W. Heparin resistance in COVID-19 patients in the intensive care unit. J Thromb Thrombolysis. 2020 Aug;50(2):287-291. doi: 10.1007/s11239-020-02145-0. PMID 32445064